CLINICAL TRIAL: NCT05537194
Title: Effects of Dihydropyridine Calcium Channel Inhibitors on Respiratory Gas Exchanges in the Intensive Care Unit: a Pharmacovigilance Study in VigiBase® and a Comparison With Urapidil
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20220908
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hypoxia
  Interventions: Drug: dihydropyridine calcium channel inhibitors use
- Patients without hypoxia
  Interventions: Drug: dihydropyridine calcium channel inhibitors use

INTERVENTIONS:
Drug: dihydropyridine calcium channel inhibitors use — administration of dihydropyridine calcium channel inhibitors

SUMMARY:
Due to their effects on hypoxic pulmonary vasoconstriction (HPV), dihydropyridine calcium channel inhibitors (CCI) could lead to hypoxia in patients with a pulmonary shunt. To the present time only preclinical studies and case reports focused on this potential adverse drug reaction. We aimed to assess the reporting association between CCI and hypoxia using the World Health Organization pharmacovigilance database (VigiBase®).

ELIGIBILITY:
Inclusion Criteria:

* present in the database

Exclusion Criteria:

* chronology not compatible with the drug imputability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Reports in VigiBase
Sampling Method: Non-Probability Sample
Enrollment: 32000000 (Actual)
Dates: Start 1963-01-01 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
association between dihydropyridine CCI or urapidil and hypoxia | from the 01/01/1963 to the 14/08/2022

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided